CLINICAL TRIAL: NCT00891020
Title: Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of Tocilizumab in Patients With Active Rheumatoid Arthritis on Background Non-biologic DMARDs and Monotherapy Who Have an Inadequate Response to Current Non-Biologic or Biologic DMARDs
Brief Title: A Study Of Tocilizumab in Patients With Moderate to Severe Active Rheumatoid Arthritis Who Have an Inadequate Response to or Are Unable to Tolerate Biologic and Non-Biologic Disease-modifying Antirheumatic Drugs (DMARDs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22533
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Results first posted 2012-04-17 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (3):
- Tocilizumab 8 mg/kg Monotherapy (Experimental): Participants received Tocilizumab 8 mg/kg as a 60 minute intravenous infusion every 4 weeks for a total of 6 infusions for 24 weeks. Participants who completed the 24 week treatment period were offered the option of entering a long-term extension phase at the investigator's discretion.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]
- Tocilizumab 4 mg/kg + DMARD (Experimental): Participants received Tocilizumab (TCZ) 4 mg/kg as a 60 minute intravenous infusion every 4 weeks for a total of 6 infusions plus non-biologic disease-modifying antirheumatic drug (DMARD) of the investigator's choice for 24 weeks. Participants not achieving a 20% improvement from baseline in tender and swollen joint counts at Week 8 were to have their dosage increased to 8 mg/kg, per protocol. Beginning at Week 12 dosage increase to 8 mg/kg was at the discretion of the investigator. Participants who completed the 24 week treatment period were offered the option of entering a long-term extension phase at the investigator's discretion.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Nonbiologic DMARDs of investigator's choice
- Tocilizumab 8 mg/kg + DMARD (Experimental): Participants received Tocilizumab (TCZ) 8 mg/kg as a 60 minute intravenous infusion every 4 weeks for a total of 6 infusions plus non-biologic disease-modifying antirheumatic drug (DMARD) of the investigator's choice for 24 weeks. Participants who completed the 24 week treatment period were offered the option of entering a long-term extension phase at the investigator's discretion.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Nonbiologic DMARDs of investigator's choice

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenous every 4 weeks for 24 weeks
Drug: tocilizumab [RoActemra/Actemra] — 4 mg/kg every 4 weeks for 24 weeks
  Arms: Tocilizumab 4 mg/kg + DMARD
Drug: Nonbiologic DMARDs of investigator's choice — Nonbiologic disease-modifying antirheumatic drugs (DMARDs) As prescribed
  Arms: Tocilizumab 4 mg/kg + DMARD; Tocilizumab 8 mg/kg + DMARD

SUMMARY:
This 3 arm randomized open label study will evaluate the safety, tolerability and efficacy of tocilizumab in patients with moderate to severe active rheumatoid arthritis, who have had inadequate response to or are unable to tolerate DMARDs. The protocol incorporates risk mitigation strategies developed in partnership with the FDA to manage known and potential risks associated with the treatment of tocilizumab. Patients will be randomized to receive tocilizumab either 4 mg/kg intravenous (iv) or 8 mg/kg iv with concomitant non-biologic DMARDs, or 8 mg/kg iv without concomitant non-biologic DMARDs, every 4 weeks, for a total of 6 infusions. The anticipated time on study treatment is 3-12 months, and the target sample size is 500-1000 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* moderate to severe active rheumatoid arthritis for >6 months;
* inadequate clinical response or unable to tolerate current or prior biologic or non-biologic Disease-modifying antirheumatic drug (DMARD) therapy;
* Swollen joint count (SJC) >/=4 and Tender joint count (TJC) >/=4
* body weight </=150kg
* current permitted non-biologic DMARDs must be on stable dose for >/= 7 weeks prior to baseline;

Exclusion Criteria:

* history of autoimmune disease or inflammatory joint disease other than rheumatoid arthritis;
* functional class IV as defined by the American College of Rheumatology (ACR) Classification of Functional Status in rheumatoid arthritis;
* treatment with rituximab within 6 months before screening;
* intraarticular corticosteroids within 8 weeks or intramuscular (im)/ intravenous (iv) corticosteroids within 12 weeks prior to screening;
* known active current or history of recurrent infections, or any major episode of infection requiring hospitalization or treatment with iv antibiotics within 4 weeks of screening, or oral antibiotics within 2 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 886 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (204):
- United States (204):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Tuscaloosa, Alabama
  - Hot Springs, Arizona
  - Paradise Valley, Arizona
  - Peoria, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Fayetteville, Arkansas
  - Fort Smith, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Covina, California
  - Escondido, California
  - Fullerton, California
  - Huntington Beach, California
  - La Jolla, California
  - Lakewood, California
  - Long Beach, California
  - Los Angeles, California
  - Murrieta, California
  - Newport Beach, California
  - Pasadena, California
  - Sacramento, California
  - San Diego, California
  - San Leandro, California
  - Santa Barbara, California
  - Santa Maria, California
  - Sherman Oaks, California
  - Van Nuys, California
  - Victorville, California
  - Westlake Village, California
  - Whittier, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Bridgeport, Connecticut
  - Danbury, Connecticut
  - Hamden, Connecticut
  - Trumbull, Connecticut
  - Lewes, Delaware
  - Aventura, Florida
  - Boca Raton, Florida
  - Clearwater, Florida
  - Dunedin, Florida
  - Fort Lauderdale, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Lake Mary, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Naples, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Gainesville, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Nampa, Idaho
  - Chicago, Illinois
  - Maywood, Illinois
  - Moline, Illinois
  - Morton Grove, Illinois
  - Peoria, Illinois
  - Schaumburg, Illinois
  - Springfield, Illinois
  - Vernon Hills, Illinois
  - Evansville, Indiana
  - Fort Wayne, Indiana
  - South Bend, Indiana
  - Cedar Rapids, Iowa
  - Lees Summit, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Monroe, Louisiana
  - New Orleans, Louisiana
  - Columbia, Maryland
  - Ellicott City, Maryland
  - Frederick, Maryland
  - Wheaton, Maryland
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Pascagoula, Massachusetts
  - Peabody, Massachusetts
  - Plymouth, Massachusetts
  - Worcester, Massachusetts
  - Battle Creek, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Petoskey, Michigan
  - Saint Clair Shores, Michigan
  - Duluth, Minnesota
  - Eagan, Minnesota
  - Edina, Minnesota
  - Saint Louis Park, Minnesota
  - Flowood, Mississippi
  - Hattiesburg, Mississippi
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - Florissant, Missouri
  - St Louis, Missouri
  - Kalispell, Montana
  - Grand Island, Nebraska
  - Lincoln, Nebraska
  - Reno, Nevada
  - Dover, New Hampshire
  - Lebanon, New Hampshire
  - Clifton, New Jersey
  - Haddon Heights, New Jersey
  - Manalapan, New Jersey
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Trenton, New Jersey
  - Voorhees Township, New Jersey
  - Las Cruces, New Mexico
  - Albany, New York
  - Binghamton, New York
  - Brooklyn, New York
  - Cooperstown, New York
  - Hewlett, New York
  - Lake Success, New York
  - New York, New York
  - Olean, New York
  - Orchard Park, New York
  - Plainview, New York
  - Rochester, New York
  - Roslyn, New York
  - Smithtown, New York
  - Syracuse, New York
  - Utica, New York
  - Asheville, North Carolina
  - Belmont, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Rock Hill, North Carolina
  - Wilmington, North Carolina
  - Bismarck, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Gallipolis, Ohio
  - Mayfield, Ohio
  - Middleburg Heights, Ohio
  - Perryburg, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Lake Oswego, Oregon
  - Bethlehem, Pennsylvania
  - Camp Hill, Pennsylvania
  - Duncansville, Pennsylvania
  - Lebanon, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pottstown, Pennsylvania
  - West Reading, Pennsylvania
  - Wexford, Pennsylvania
  - Willow Grove, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Hickory Grove, South Carolina
  - Myrtle Beach, South Carolina
  - Hendersonville, Tennessee
  - Hixson, Tennessee
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Mesquite, Texas
  - Nassau Bay, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Waco, Texas
  - Burlington, Vermont
  - Arlington, Virginia
  - Burke, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Olympia, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Beckley, West Virginia
  - Clarksburg, West Virginia
  - Brookfield, Wisconsin
  - Franklin, Wisconsin
  - Glendale, Wisconsin
  - Milwaukee, Wisconsin
  - Onalaska, Wisconsin

REFERENCES:
- [Derived] Weinblatt ME, Kremer J, Cush J, Rigby W, Teng LL, Devenport J, Singh N, Lepley D, Genovese MC. Tocilizumab as monotherapy or in combination with nonbiologic disease-modifying antirheumatic drugs: twenty-four-week results of an open-label, clinical practice study. Arthritis Care Res (Hoboken). 2013 Mar;65(3):362-71. doi: 10.1002/acr.21847. PMID 22972745

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1129 patients were screened for the study. Of these 1129 patients, 886 patients were enrolled and 243 patients were screen failures.
Groups:
- Tocilizumab 8 mg/kg Monotherapy: Participants received Tocilizumab 8 mg/kg as a 60 minute intravenous infusion every 4 weeks for a total of 6 infusions for 24 weeks. Participants who completed the 24 week treatment period were offered the option of entering a long-term extension phase.
- Tocilizumab 4 mg/kg + DMARD: Participants received Tocilizumab (TCZ) 4 mg/kg as a 60 minute intravenous infusion every 4 weeks for a total of 6 infusion plus non-biologic disease-modifying antirheumatic drug (DMARD) of the investigator's choice for 24 weeks. Participants not achieving a 20% improvement from baseline in tender and swollen joint counts at Week 8 were to have their dosage increased to 8 mg/kg, per protocol. Beginning at Week 12 dosage increase to 8 mg/kg was at the discretion of the investigator. Participants who completed the 24 week treatment period were offered the option of entering a long-term extension phase.
- Tocilizumab 8 mg/kg + DMARD: Participants received Tocilizumab 8 mg/kg as a 60 minute intravenous infusion every 4 weeks for a total of 6 infusion plus non-biologic disease-modifying antirheumatic drug (DMARD) of the investigator's choice for 24 weeks. The dosage could be decreased to 4 mg/kg for safety reasons at the investigator's discretion. Participants who completed the 24 week treatment period were offered the option of entering a long-term extension phase.
Period: 24 Week Treatment Period
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Started | 163 | 363 | 360
Intent-to-Treat (ITT) | 163 | 362 | 358
Safety Set | 138 (4 patients from 8 mg/kg +DMARD arm did not receive DMARD, included in Monotherapy arm for safety.) | 364 (1 patient from Monotherapy arm and 1 from 8 mg/kg +DMARD, included in 4 mg/kg +DMARD arm for safety.) | 381 (28 patients from Monotherapy arm received DMARD, included in 8 mg/kg +DMARD arm for safety.)
Completed | 126 | 303 | 302
Not Completed | 37 | 60 | 58
Not completed — Adverse event or intercurrent illness | 11 | 32 | 17
Not completed — Death | 0 | 2 | 0
Not completed — Insufficient therapeutic response | 6 | 9 | 15
Not completed — Failure to return | 4 | 5 | 5
Not completed — Violation of selection criteria at entry | 1 | 0 | 2
Not completed — Other protocol violation | 1 | 1 | 2
Not completed — Refused treatment/did not cooperate | 3 | 2 | 1
Not completed — Withdrew consent | 6 | 3 | 15
Not completed — Administrative/Other | 5 | 6 | 1
Period: Long-term Extension Period
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Started | 55 | 196 | 193
Completed | 49 | 172 | 170
Not Completed | 6 | 24 | 23
Not completed — Adverse Event | 1 | 11 | 10
Not completed — Death | 0 | 0 | 1
Not completed — Insufficient therapeutic response | 3 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Refused treatment/did not cooperate | 1 | 6 | 4
Not completed — Failure to return | 0 | 2 | 3
Not completed — Administrative | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD | Total
Number analyzed (Participants) | 138 | 364 | 381 | 883
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measures are based on the number of participants in the Safety Population who received at least one dose of study drug and who had at least one post baseline safety assessment.
  years | 53.5 (12.63) | 55.6 (11.92) | 54.0 (12.11) | 54.6 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 273 | 296 | 679
  Male | 28 | 91 | 85 | 204

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing at Least One Serious Adverse Event (SAE) During the 24 Week Treatment Period
Description: An SAE was any adverse event that at any dose fulfilled at least one of the following criteria:
  * Was fatal (results in death)
  * Was life-threatening
  * Required in-patient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was medically significant or required intervention to prevent one or other of the outcomes listed above.
Time Frame: 24 Weeks
Population: Safety Population. Patients were included in the TCZ dose group according to the first infusion they actually received. Patients were assigned as using a nonbiologic DMARD if they took at least 1 dose of nonbiologic DMARD during the treatment period. Patients who did not take at least 1 dose of nonbiologic DMARD were considered as on monotherapy.
Measure: Number; unit: Percentage of Participants
Groups:
- Tocilizumab 8 mg/kg Monotherapy: Participants received Tocilizumab (TCZ) 8 mg/kg as a 60 minute intravenous infusion every 4 weeks for a total of 6 infusions for 24 weeks. Participants who completed the 24 week treatment period were offered the option of entering a long-term extension phase.
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Number analyzed (Participants) | 138 | 364 | 381
Percentage of Participants | 5.8 | 8.0 | 8.4

2. Secondary Outcome: Percentage of Participants Experiencing Serious Adverse Events of Special Interest
Description: Serious Adverse Events of Special interest include:
  * Serious infections including opportunistic infections
  * Complications of diverticulitis (including lower gastrointestinal [GI] perforations)
  * Myocardial infarction/acute coronary syndrome
  * Stroke
  * Spontaneous or serious bleeding
  * Malignant neoplasms
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Number analyzed (Participants) | 138 | 364 | 381
Percentage of Participants
  Serious Infections (including opportunistic) | 2.9 | 3.6 | 3.9
  Gastrointestinal Perforations and Related Events | 0 | 0.8 | 0
  Myocardial Infarction/Acute Coronary Syndrome | 0 | 0 | 0.3
  Stroke | 0 | 0.3 | 0
  Spontaneous/Serious Bleeding | 0 | 0.3 | 0.3
  Malignant Neoplasms | 0 | 0 | 0.3

3. Secondary Outcome: Percentage of Participants Experiencing Non-serious Adverse Events of Special Interest
Description: Non-serious adverse Events of Special interest include:
  * Serious/Medically Significant Hepatic Events
  * Spontaneous /Serious Bleeding
  * Malignant Neoplasms
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Number analyzed (Participants) | 138 | 364 | 381
Percentage of Participants
  Serious/Medically Significant Hepatic Events | 0 | 0 | 0.3
  Spontaneous/Serious Bleeding | 4.3 | 3.3 | 7.3
  Malignant Neoplasms | 0 | 0.3 | 0.3

4. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Weeks 8, 16, and 24
Description: Clinical Remission is defined as a Disease Activity Score 28 [DAS28] < 2.6. The DAS28 is a combined index for measuring disease activity in RA. The index includes tender joint count (TJC) -28 joints and swollen joint count (SJC)-28 joints, acute phase response (CRP) and general health status. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Weeks 8,16,24
Population: Intent-to-treat population includes participants who received at least one dose of study drug. Patients were included in the treatment group to which they were randomized or assigned, regardless of the treatment actually received. "n" in each of the categories is the number of participants with data available for analysis at the given time point.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Number analyzed (Participants) | 163 | 362 | 358
Percentage of Participants
  Week 8 (n=147, 337, 334) | 8.8 | 6.8 | 12.9
  Week 16 (n=127, 317, 304) | 15.7 | 17.4 | 22.0
  Week 24 (n=126, 286, 302) | 19.8 | 20.6 | 25.2

5. Secondary Outcome: Change From Baseline in DAS28 Score at Weeks 8, 16 and 24
Description: The DAS28 is a combined index for measuring disease activity in rheumatoid arthritis (RA). The index includes tender joint count (TJC) -28 joints and swollen joint count (SJC)-28 joints, acute phase response C-reactive protein (CRP) and general health status. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A score of < 2.6 represents clinical remission, a score of ≤ 3.2 represents low disease activity, and a score of > 5.1 represents high disease activity.
  The Change from Baseline to Weeks 8, 16 and 24 is reported.
Time Frame: Baseline, Weeks 8,16,24
Population: Intent-to-treat includes participants who received at least one dose of study drug. Patients were included in the treatment group to which they were randomized or assigned, regardless of the treatment actually received. "n" in each of the categories is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Number analyzed (Participants) | 163 | 362 | 358
Score on a scale
  Week 8 (n=147, 337, 334) | -1.75 (1.213) | -1.00 (1.189) | -1.54 (1.187)
  Week 16 (n=127, 317, 304) | -2.07 (1.406) | -1.66 (1.244) | -1.87 (1.322)
  Week 24 (n=126, 286, 302) | -2.03 (1.384) | -1.81 (1.264) | -1.94 (1.380)

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) (ACR20/50/70) Responses at Weeks 8, 16, and 24
Description: The ACR response rates ACR20, ACR50, and ACR70 are defined as ≥20%, ≥50%, and ≥70% improvement from baseline, respectively, in:
  1. Swollen Joint Count (66 joints) and Tender Joint Count (68 joints) and
  2. At least 3 of the following 5 assessments:
     * Patient's global assessment of pain-Visual Analog Scale (VAS)
     * Patient global assessment of disease activity-(VAS)
     * Physician global assessment of disease activity-(VAS)
     * Patient assessment of disability (physical function scale of the Multidimensional Health Assessment Questionnaire)
     * Acute phase response C-Reactive Protein (CRP)
Time Frame: Baseline, Weeks 8,16,24
Population: Intent-to-treat population includes all participants who received at least one dose of study drug. Patients were included in the treatment group to which they were randomized or assigned, regardless of the treatment actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Number analyzed (Participants) | 163 | 362 | 358
Percentage of Participants
  Week 8 ACR20 responders | 40.5 | 37.8 | 40.8
  Week 8 ACR50 responders | 14.7 | 11.9 | 16.8
  Week 8 ACR70 responders | 4.3 | 3.3 | 5.6
  Week 16 ACR20 responders | 46.6 | 43.9 | 45.3
  Week 16 ACR50 responders | 23.3 | 19.9 | 22.3
  Week 16 ACR70 responders | 7.4 | 8.6 | 9.8
  Week 24 ACR20 responders | 47.9 | 44.8 | 49.7
  Week 24 ACR50 responders | 24.5 | 24.3 | 27.1
  Week 24 ACR70 responders | 7.4 | 8.8 | 10.3

7. Secondary Outcome: Percentage of Participants With Tocilizumab Dose Increased From 4 mg/kg to 8 mg/kg at Week 8
Description: Dosage could be increased from 4 mg/kg Tocilizumab to 8 mg/kg due to failure to achieve 20% improvement from baseline in swollen and tender joint counts.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab 4 mg/kg + DMARD
Number analyzed (Participants) | 364
Percentage of Participants | 39.9

8. Secondary Outcome: Number of Participants Having Their Tocilizumab Dose Increased From 4 mg/kg to 8 mg/kg at Weeks 12, 16, and 20
Description: Dosage of Tocilizumab 4 mg/kg could be increased to 8 mg/kg at the discretion of the investigator based on assessment of the patient's benefit-risk after Week 12.
Time Frame: Weeks 12,16, 20
Population: Safety population includes participants who received at least one dose of study drug. "n" in each of the categories is the number of participants previously on 4mg/kg + DMARD and receiving a dose at the current visit. Patients were assigned as using a nonbiologic DMARD if they took at least 1 dose of nonbiologic DMARD during the treatment period.
Measure: Number; unit: Participants
Arm/Group | Tocilizumab 4 mg/kg + DMARD
Number analyzed (Participants) | 364
Participants
  Week 12 (n=183) | 41
  Week 16 (n=138) | 18
  Week 20 (n=119) | 5

9. Secondary Outcome: Change From Baseline in Routine Assessment Patient Index Data (RAPID3) Score at Weeks 8, 16, and 24
Description: The RAPID3 is a combined index derived from the Multidimensional Health Assessment Questionnaire that includes physical function score, pain Visual Analog Scale (VAS), and global assessment of disease activity VAS. The total RAPID3 score ranges from 0 to 10 where higher scores represent worse outcomes. A negative change from baseline indicates improvement.
Time Frame: Baseline, Weeks 8,16,24
Population: Intent-to-treat population includes all participants who received at least 1 dose of study drug. Patients were included in the treatment group to which they were randomized or assigned, regardless of the treatment actually received. "n" in each of the categories is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Number analyzed (Participants) | 163 | 362 | 358
Score on a scale
  Week 8 (n=156, 348, 343) | -1.60 (1.803) | -1.10 (1.848) | -1.28 (1.733)
  Week 16 (n=138, 325, 315) | -1.97 (2.068) | -1.42 (1.896) | -1.46 (1.897)
  Week 24 (n=134, 306, 308) | -1.83 (1.978) | -1.61 (1.972) | -1.46 (1.962)

10. Secondary Outcome: Change From Baseline in Fatigue Visual Analogue Scale (VAS) at Weeks 8, 16, and 24
Description: The fatigue VAS is a single-item, patient-reported outcome that measures the severity of the fatigue over the past week. Patients rate their fatigue on a scale of 0 (fatigue is no problem) to 100 (fatigue is a major problem). Higher scores represent higher disease activity and a negative change from baseline indicates improvement.
Time Frame: Baseline, Weeks 8,16,24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Number analyzed (Participants) | 163 | 362 | 358
Score on a scale
  Week 8 (n=156, 350, 344) | -13.17 (25.584) | -10.06 (25.349) | -13.33 (24.950)
  Week 16 (n=138, 329, 317) | -19.38 (26.639) | -14.00 (26.282) | -15.58 (25.802)
  Week 24 (n=135, 307, 312) | -15.85 (26.881) | -16.73 (26.261) | -16.07 (26.321)

ADVERSE EVENTS:
Time Frame: Includes Adverse Events that occurred during the 24-week Treatment Period and the Long-term Extension Period (up to 72 Weeks)
Description: Safety population. Patients were included in the TCZ dose group according to the first infusion they actually received. Patients were assigned as using a nonbiologic DMARD if they took at least 1 dose of nonbiologic DMARD during the treatment period. Patients who did not take at least 1 dose of nonbiologic DMARD were considered as on monotherapy.
Arm/Group | Tocilizumab 8 mg/kg Monotherapy | Tocilizumab 4 mg/kg + DMARD | Tocilizumab 8 mg/kg + DMARD
Serious Adverse Events (participants affected / at risk) | 11/138 | 45/364 | 40/381
Other Adverse Events (participants affected / at risk) | 63/138 | 185/364 | 189/381
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg Monotherapy (N=138) | Tocilizumab 4 mg/kg + DMARD (N=364) | Tocilizumab 8 mg/kg + DMARD (N=381)
Pneumonia (Infections and infestations) | 1 | 5 | 8
Cellulitis (Infections and infestations) | 2 | 6 | 3
Osteomyelitis (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2
Abscess intestinal (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 1 | 1
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 3 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Vesical fistula (Renal and urinary disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pyothorax (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac valve rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg Monotherapy (N=138) | Tocilizumab 4 mg/kg + DMARD (N=364) | Tocilizumab 8 mg/kg + DMARD (N=381)
Upper respiratory tract infection (Infections and infestations) | 14 | 36 | 41
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 12 | 40 | 32
Sinusitis (Infections and infestations) | 11 | 33 | 36
Headache (Nervous system disorders) | 7 | 27 | 26
Nasopharyngitis (Infections and infestations) | 7 | 31 | 19
Diarrhoea (Gastrointestinal disorders) | 9 | 25 | 14
Alanine aminotransferase increased (Investigations) | 8 | 13 | 26
Rash (Skin and subcutaneous tissue disorders) | 4 | 13 | 23
Urinary tract infection (Infections and infestations) | 8 | 8 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 20 | 22
Nausea (Gastrointestinal disorders) | 5 | 25 | 16
Chest pain (General disorders) | 7 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.